CLINICAL TRIAL: NCT00880152
Title: Mindfulness-Based Stress Reduction for Posttraumatic Stress Disorder: A Pilot Study
Brief Title: Mindfulness Based Stress Reduction for Posttraumatic Stress Disorder: A Pilot Study
Acronym: MBSRforPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Puget Sound Partners for Global Health (Unknown)
Responsible Party: David Kearney, M.D., VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34622
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Stress Disorders, Post-Traumatic; Depression
Keywords: stress; mindfulness; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Wounds and Injuries | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBSR (Experimental): An 8-week course in mindfulness-based stress reduction (MBSR)
  Interventions: Behavioral: Mindfulness-based stress reduction
- 2 (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — An 8-week course in mindfulness training
  Arms: MBSR

SUMMARY:
PTSD is a common consequence of war, for soldiers and civilians. PTSD results in hyperarousal, avoidance, numbing, and re-experiencing, causing persistent decreased quality of life. Mindfulness involves the ability to bring attention to the present moment without judgment; this ability is correlated with measures of mental health. Within health care, mindfulness is taught as an 8-week course called Mindfulness-Based Stress Reduction (MBSR). MBSR is unstudied for PTSD. We propose to assess the feasibility of MBSR as an intervention for PTSD, since it may affect hypervigilance, avoidance, and reactivity associated with this disorder.

Specific Aims: Aim 1: Assess the feasibility of recruiting and retaining a sample of veterans with PTSD to complete a study protocol that involves randomization to usual care or usual care plus MBSR. Aim 2: Apply measures of PTSD symptom severity, depression and quality of life before and after randomization, to assess whether there is evidence of benefit and whether MBSR warrants further study for PTSD, and allow calculation of standardized effect sizes. Aim 3: Apply a validated measure of mindfulness before and after treatment. Aim 4: Explore the relationship between PTSD symptoms, mindfulness score, and frequency of meditation practice.

ELIGIBILITY:
Inclusion Criteria:

* Must have PTSD

Exclusion Criteria:

* Active substance use
* Active suicidal ideations
* Borderline or antisocial personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
PTSD symptom score | baseline, after MBSR and 4 months later

SECONDARY OUTCOMES:
depression (PHQ9) | baseline, after MBSR and 4 months later

CONTACTS AND LOCATIONS:
Overall Officials: David Kearney, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Derived] Kearney DJ, McDermott K, Malte C, Martinez M, Simpson TL. Effects of participation in a mindfulness program for veterans with posttraumatic stress disorder: a randomized controlled pilot study. J Clin Psychol. 2013 Jan;69(1):14-27. doi: 10.1002/jclp.21911. Epub 2012 Aug 28. PMID 22930491